CLINICAL TRIAL: NCT00251173
Title: Services Interventions for Injured ED Substance Abusers
Brief Title: Project Health Link: Connecting Patients With Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Frederic C. Blow, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01DA016591-01A1 (NIH)
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strengths Based Case Management Model (SBCM) (Active Comparator): The Strengths Based Case Management Model (SBCM) consists of 5 case-management sessions designed to promote linkage and engagement in assessment and treatment services, while assisting with the patient's perceived needs, as well as personal strengths and barriers to linkage and engagement.
  Interventions: Behavioral: Strengths Based Case Management (SBCM)
- Motivational Enhancement Therapy (MET) (Active Comparator): The MET therapist will conduct 2 motivational enhancement sessions to work through the content of an educational workbook targeting the participant's substance use/abuse with the goal of negotiating a 'contract' to: 1) link to services, with the eventual goal of seeking and receiving specialized substance treatment; or 2) provide a strategy to self-monitor substance use, consider consequences, and later seek assessment.
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)
- Brief Informational Feedback (BIF) session (Active Comparator): Subjects will receive brief informational feedback on the results of their alcohol screening and assessment and encouragement to seek treatment.
  Interventions: Behavioral: Brief Informational Feedback (BIF) session

INTERVENTIONS:
Behavioral: Strengths Based Case Management (SBCM)
  Arms: Strengths Based Case Management Model (SBCM)
Behavioral: Motivational Enhancement Therapy (MET)
  Arms: Motivational Enhancement Therapy (MET)
Behavioral: Brief Informational Feedback (BIF) session
  Arms: Brief Informational Feedback (BIF) session

SUMMARY:
The proposed study will compare three alternative interventions in the emergency department (ED) to promote linkage to substance abuse assessment, referral and treatment entry for those who meet abuse/dependence criteria for stimulants, cannabis, and/or non-injected opioids: (1) a 5-session Strengths-Based Case Management (SBCM) model; (2) a 2-session Brief Motivational Enhancement (BME); or (3) a one-time Brief Informational Feedback (BIF) session. The primary outcome variables for this trial include receiving an assessment and referral and treatment entry. Other outcomes include degree of treatment completion, substance-related measures, health service utilization, health status changes, and psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* (1) adults age 19-60 presenting to the Hurley Medical Center ED within 24 hours of an injury; (2) ability to provide informed consent.

Additional inclusion criteria for intervention study: meets criteria for substance abuse or dependence for stimulants (cocaine powder, crack cocaine, methamphetamine, amphetamine), cannabis (marijuana, hashish), and or opioids (noninjected heroin, other opioids such as hydrocodone and oxycodone) in the previous year.

Exclusion Criteria:

* (1) adult patients who do not understand English; (2) prisoners; (3) adults classified by medical staff as "Level 1 trauma"; (4) adults deemed unable to provide informed consent as stated above (e.g., intoxication, mental incompetence); (5) patients treated in the ED for suicide attempts and sexual assaults; (6) patients who have been in treatment for substance abuse in the past six months; (7) patients who are triaged to psychiatric emergency services; and (8) patients who report injecting heroin or other opiates in the past year.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 755 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
receipt of assessment | 3 and 6 months post-baseline
treatment entry | 3 and 6 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No